CLINICAL TRIAL: NCT02489695
Title: Multicenter Phase II Study of Axitinib in First Line Treatment for Patients With Locally Advanced or Metastatic Papillary Renal Cell Carcinoma (PRCC)
Brief Title: Axitinib in1st Line Treatment for Patients With Advanced or Metastatic Papillary Renal Cell Carcinoma
Acronym: AXIPAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXIPAP; ET14-090 (Other: Centre Léon Bérard)
Record Dates: First submitted 2015-06-19; First posted 2015-07-03 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Papillary Renal Cell Carcinoma
Keywords: locally advanced or metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- axitinib + pembrolizumab (Experimental): axitinib 10mg twice a day
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — axitinib 10mg twice a day

SUMMARY:
Multicenter, single arm, phase II study using a A'Hern single-stage procedure in patients with locally advanced or metastatic papillary renal cell carcinoma (PRCC) in first-line treatment.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) accounts for 2-3% of all adult malignancies worldwide, representing the seventh most common cancer in men and the ninth in women. The annual incidence is more than 337 000 cases and around 140 000 persons die every year. Half of patients with RCC are going to develop metastases, either with synchronous metastatic sites (25%) or during the follow up (25%).

Papillary renal cell carcinoma (PRCC) represents 10-15% of RCC and is characterized by a cytogenetic profile distinct from other types of renal cancer. Histologically, PRCC could be separated in 2 distinct subtypes: type 1 and type 2.

Vascular endothelial growth factor (VEGF) is a potent induction factor, playing a central role in angiogenesis and vascular permeability of tumor tissues. It binds to three specific receptors: VEGFR-1, VEGFR-2 and VEGFR-3, which are thus implicated in pathologic angiogenesis, tumor growth and metastatic progression of cancer. Patients with papillary histology demonstrated high expression of VEGF and VEGFR-2, making VEGF-targeted therapy an attractive therapeutic option.

Recently, several studies have been developed to assess VEGF targeted therapy in patients with PRCC, mostly with sunitinib and with poor results (median progression-free survival (PFS) around 6 months).

Axitinib is a potent, selective second-generation inhibitor of all three VEGF receptors. By inhibiting VEGF-mediated endothelial cell proliferation and survival, axitinib inhibits angiogenesis and tumor growth.

In phase II trials, axitinib has shown anti-tumor activity with well-tolerated clinical safety profile in patients with advanced solid tumors, including RCC.

Axitinib has been approved for the second-line treatment of advanced RCC on the basis of the pivotal randomized phase III AXIS trial results. 723 patients were enrolled and randomly assigned to receive axitinib or sorafenib. The median PFS assessed by independent review committee was 6.7 months with axitinib compared to 4.7 months with sorafenib (hazard ratio 0.665; 95% CI 0.544-0.812; one-sided p<0.0001).

In all studies, the safety analysis showed a good tolerance of axitinib. The most common adverse reactions (occurring in >20% of treated subjects) were diarrhea, hypertension, fatigue, decreased appetite, nausea, dysphonia and hand-foot skin reaction. Dose discontinuations were reported in 4% of patients with axitinib vs. 8% with sorafenib.

Little clinical data regarding the efficacy of recently developed VEGF targeted therapies in first-line treatment of PRCC is available. To date, there is no standard treatment, and evaluation of efficacy of the new targeted agents is clearly needed.

The purpose of this study is to evaluate the efficacy and safety of axitinib in first-line treatment of patients with papillary renal cell carcinoma.

Axitinib inhibits angiogenesis and vascular permeability in tumor tissues, leading to inhibition of tumor growth.

Axitinib has shown antitumor activity in patients with RCC in phase II and III clinical trials.

VEGF inhibitors are currently used in PRCC treatment, with disappointing results. Axitinib is more potent and selective against the VEGFR family compared with sorafenib and sunitinib in biochemical assays, and could have a similar efficacy with lesser toxicities, therefore may provide a clinical benefit in patients with PRCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Metastatic or locally advanced (inoperable) pure type 1 or 2 or mixed PRCC, histologically confirmed by central review: relevant slides [and blocks if available] with the initial histology report must be sent for central reading before confirmation of inclusion.
3. No prior systemic treatment for metastatic renal cancer (chemotherapy, immunotherapy, anti-angiogenic drugs, or treatment under evaluation).
4. At least one measurable site of disease as defined by RECIST 1.1 criteria.
5. ECOG performance status of 0, 1.
6. No toxicity > 1 according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
7. In case of prior radiation therapy, discontinuation of irradiation for at least 4 weeks before first dose of study treatment. This period can be reduced to at least 1 week in case of radiotherapy in a limited field (< 10% of the whole body) while no side effects grade ≥ 2 is expected and keeping at least one site for evaluation.
8. Adequate bone marrow, liver and renal function, as defined below:

   * Absolute neutrophil count ≥ 1.5 G/L, platelet count ≥ 100 G/L, and hemoglobin ≥ 9 g/dL),
   * AST/ALT ≤ 3 x upper limit of normal (ULN) (or ≤ 5.0 x ULN if liver metastasis) and total bilirubin ≤ 1.5 x ULN (≤ 2.5 x ULN if liver metastases),
   * Serum creatinine ≤ 2.0 x ULN or creatinine clearance ≥ 50 mL/min according to Cockroft formula or MDRD formula for patients older than 65 years,
9. Absence of proteinuria confirmed by urinary dipstick test. If the dipstick test is ≥ 2+, proteinuria will be quantitated on a complete 24h urine sample (< 1 g/L of protein/24h sample).
10. Adequate contraceptive methods for fertile female subjects for the whole duration of the study and for 7 days after the last dose of study drug.

    Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study.
11. Covered by a medical insurance, in countries where applicable.
12. Written informed consent before any study specific procedures or assessments.

Exclusion Criteria:

1. Prior TKI treatment in adjuvant situation for renal cancer.
2. Significant cardiovascular disease including:

   * Disorder of left ventricular function with a LVEF < 50%,
   * Uncontrolled arterial hypertension under adapted medication: systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg or both despite appropriate therapy, or patients under 3 antihypertensive therapies at screening,
   * Myocardial infarction, severe angina, or unstable angina within 6 months prior to inclusion,
   * History of serious ventricular arrhythmia (ie ventricular tachycardia or ventricular fibrillation),
   * Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication),
   * Coronary or peripheral artery bypass graft within 6 months of screening.
3. Presence of brain metastases on MRI or CT-scan performed within 28 days prior to inclusion. Patients with a history of brain metastases treated by surgery or stereotactic surgery, with normal brain MRI or CT-scan are allowed to participate.
4. Major surgical procedure, open biopsy, or serious none healing wound within 28 days prior to inclusion.
5. Any active acute or chronic or uncontrolled infection/disorder that impair the ability to evaluate the patient or the ability for the patient to complete the study.
6. Prior history of other malignancies other than PRCC (except for curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix) unless the subjects has been free of the disease for at least 3 years.
7. Inability to swallow oral medications, or presence of active inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhea.
8. Patient included in another clinical trial, except for supportive care trials.
9. Psychological, familial, sociological, or geographical conditions that would limit compliance with study protocol requirements.
10. Pregnant or breastfeeding women (mandatory negative serum or urinary pregnancy test at study entry for all women of childbearing potential).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
The efficacy of axitinib in first-line treatment of PRCC. | 24-week
  24-week progression-free rate

SECONDARY OUTCOMES:
The safety of axitinib in patients with PRCC (NCI CTCAE v4) | Week 2, 4, 8, 16 then Month 4, 6, 8,10, 12, 14, 16,18
The progression-free survival (RECIST 1.1) in each PRCC subtypes | Week 2, 4, 8, 16 then Month 4, 6, 8,10, 12, 14, 16,18
The overall survival | 43 month after first inclusion
The best response | Week 2, 4, 8, 16 then Month 4, 6, 8,10, 12, 14, 16,18
  the best response recorded from the start of the treatment until disease progression
the objective response rate | Week 2, 4, 8, 16 then Month 4, 6, 8,10, 12, 14, 16,18
the duration of response | Week 2, 4, 8, 16 then Month 4, 6, 8,10, 12, 14, 16,18

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie NEGRIER, PhD, Principal Investigator — Centre Leon Berard
Locations (10):
- France (10):
  - ICO Paul Papin, Angers
  - Chu Bordeaux, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Geogres François Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICO - René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - ICL, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

REFERENCES:
- [Background] Negrier S, Rioux-Leclercq N, Ferlay C, Gross-Goupil M, Gravis G, Geoffrois L, Chevreau C, Boyle H, Rolland F, Blanc E, Ravaud A, Dermeche S, Flechon A, Albiges L, Perol D, Escudier B; GETUG collaborative group. Axitinib in first-line for patients with metastatic papillary renal cell carcinoma: Results of the multicentre, open-label, single-arm, phase II AXIPAP trial. Eur J Cancer. 2020 Apr;129:107-116. doi: 10.1016/j.ejca.2020.02.001. Epub 2020 Mar 5. PMID 32146304
- [Derived] de Vries-Brilland M, Rioux-Leclercq N, Meylan M, Dauve J, Passot C, Spirina-Menand E, Flippot R, Fromont G, Gravis G, Geoffrois L, Chevreau C, Rolland F, Blanc E, Lefort F, Ravaud A, Gross-Goupil M, Escudier B, Negrier S, Albiges L. Comprehensive analyses of immune tumor microenvironment in papillary renal cell carcinoma. J Immunother Cancer. 2023 Nov;11(11):e006885. doi: 10.1136/jitc-2023-006885. PMID 37935564